CLINICAL TRIAL: NCT04759560
Title: Biometric Characteristics Of The Eye With Microcornea/Microphthalmia And Congenital Cataract Before And After Cataract Extraction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Nshokano Simba Gloria, Ophthalmology resident, Alexandria University
Other Study IDs: MICROCORNEA/MICROPHTHALMIA
Record Dates: First submitted 2021-02-15; First posted 2021-02-18 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Congenital Cataract; Microphthalmos; Microcornea
Keywords: anterior segment biometry; cataract surgery; aphakia/ pseudophakia
MeSH Terms: conditions — Microphthalmos

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Early cataract surgery in microcornea/microphthalmia eyes is essential to prevent amblyopia and improve visual outcomes, including stereopsis. However, despite recent advances in pediatric cataract microsurgical techniques, this surgery remains challenging owing to several intraoperative difficulties attributable to the crowded anterior segment in these small, soft, and poorly developed eyes with shallow anterior chambers, and poor pupillary dilation.

In this study the investigator aim to report on the changes in the anterior segment biometric characteristics after cataract extraction in eyes with microcornea/microphthalmia with congenital cataract.

DETAILED DESCRIPTION:
Eyes with congenital cataract have usually small cornea due to developmental delay of the globe. Recognition of microcornea/microphthalmia may be important as a potential contributor to the development of aphakic glaucoma after cataract surgery. Biometrics characteristics of eyes with m/m before and after removal of the cataractous lens can justify the occurrence of postoperative complications, including glaucoma.

Aim of the study: to report on the changes in the anterior segment biometric characteristics after cataract extraction in eyes with microcornea/microphthalmia with congenital cataract.

Methods:

The study will be a prospective cohorte. Biometry of eligible eyes with congenital cataract in one or both eyes with horizontal cornea diameter less than 11mm and/or axial length less than 2standard deviation for age will be compare to otherwise normal eyes with congenital cataract before and after cataract extraction. The anterior segment biometric characteristics using ultrasound biomicroscopy to measure anterior chamber depth and angle.Cataract surgery will be conducted with or without intraocular lens implantation.Postoperative follow up will be scheduled at the first week and first month, third and sixth months

ELIGIBILITY:
Inclusion Criteria:

1. Children presenting with congenital cataract in one or both eyes and with a horizontal corneal diameter less than 11 mm and/or an axial length less than 2 standard deviations for age of the child, less than 18mm in children under one year and less than 20mm in those less than 1year (cases).
2. Children presenting with congenital cataract in one or both eyes with otherwise normal ocular biometric characteristics (controls).

Exclusion Criteria:

1.Children presenting with congenital cataract associated with other ocular anomalies other than microcornea/microphthalmia

Ages: 3 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All children between 3months and 7 years with congenital cataract without other ocular anomalies other than micornea/ microphthalmia; who will visit the pediatric ophthalmology clinic of Alexandria main University from july 2020 to january 2021.
Sampling Method: Non-Probability Sample
Enrollment: 133 (Estimated)
Dates: Start 2020-07-25 (Actual); Primary Completion 2021-07-25 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative changes in the biometric characteristics of eyes at 3months | 3 months
  the anterior segment biometric characteristics will be assess using ultrasound biomicroscopy
  biomicroscopy
Postoperative changes in the biometric characteristics of eyes at 6months | 6 months
  the anterior segment biometric characteristics will be assess using ultrasound biomicroscopy

SECONDARY OUTCOMES:
Postoperative complications at 3 months | 3 months
  we will report occurence of postoperative complications
Postoperative complications at 6months | 6 months
  we will report occurence of postoperative complications

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Nshokano Simba, MBBch, Principal Investigator — Alexandria University; Nader L Bayoumi, Professor, Study Director — Alexandria University; Nihal Mohamed Elshakankiri, Professor, Study Chair — Alexandria University
Locations (1):
- Faculty of Medecine, Alexandria, Alexandria/ Egypt, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Praveen MR, Vasavada AR, Shah SK, Khamar MB, Trivedi RH. Long-term postoperative outcomes after bilateral congenital cataract surgery in eyes with microphthalmos. J Cataract Refract Surg. 2015 Sep;41(9):1910-8. doi: 10.1016/j.jcrs.2015.10.005. PMID 26603400
- [Background] Ventura MC, Sampaio VV, Ventura BV, Ventura LO, Nose W. Congenital cataract surgery with intraocular lens implantation in microphthalmic eyes: visual outcomes and complications. Arq Bras Oftalmol. 2013 Jul-Aug;76(4):240-3. doi: 10.1590/s0004-27492013000400011. PMID 24061837
- [Background] Wu X, Long E, Lin H, Liu Y. Prevalence and epidemiological characteristics of congenital cataract: a systematic review and meta-analysis. Sci Rep. 2016 Jun 23;6:28564. doi: 10.1038/srep28564. PMID 27334676
- [Background] Chen D, Gong XH, Xie H, Zhu XN, Li J, Zhao YE. The long-term anterior segment configuration after pediatric cataract surgery and the association with secondary glaucoma. Sci Rep. 2017 Feb 21;7:43015. doi: 10.1038/srep43015. PMID 28220849
- [Background] Prasad S, Ram J, Sukhija J, Pandav SS, Gupta PC. Cataract surgery in infants with microphthalmos. Graefes Arch Clin Exp Ophthalmol. 2015 May;253(5):739-43. doi: 10.1007/s00417-014-2908-8. Epub 2015 Jan 16. PMID 25592478
- [Background] Khokhar SK, Dave V. Cataract surgery in infant eyes with microphthalmos. J Cataract Refract Surg. 2009 Oct;35(10):1844; author reply 1844-5. doi: 10.1016/j.jcrs.2009.05.040. No abstract available. PMID 19781495
- [Background] Vasavada VA, Dixit NV, Ravat FA, Praveen MR, Shah SK, Vasavada V, Vasavada AR, Trivedi RH. Intraoperative performance and postoperative outcomes of cataract surgery in infant eyes with microphthalmos. J Cataract Refract Surg. 2009 Mar;35(3):519-28. doi: 10.1016/j.jcrs.2008.11.031. PMID 19251147
- [Background] Filous A, Osmera J, Hlozanek M, Mahelkova G. Central corneal thickness in microphthalmic eyes with or without history of congenital cataract surgery. Eur J Ophthalmol. 2011 Jul-Aug;21(4):374-8. doi: 10.5301/EJO.2010.6090. PMID 21140367
- [Background] Nishina S, Noda E, Azuma N. Outcome of early surgery for bilateral congenital cataracts in eyes with microcornea. Am J Ophthalmol. 2007 Aug;144(2):276-280. doi: 10.1016/j.ajo.2007.04.019. Epub 2007 May 29. PMID 17533105
- [Background] Abouzeid H, Meire FM, Osman I, ElShakankiri N, Bolay S, Munier FL, Schorderet DF. A new locus for congenital cataract, microcornea, microphthalmia, and atypical iris coloboma maps to chromosome 2. Ophthalmology. 2009 Jan;116(1):154-162.e1. doi: 10.1016/j.ophtha.2008.08.044. Epub 2008 Nov 12. PMID 19004499
- [Result] Majid S, Ateeq A, Bukari S, Hussain M. Outcomes of cataract surgery in Microophthalmia. Pak J Med Sci. 2018 Nov-Dec;34(6):1525-1528. doi: 10.12669/pjms.346.14622. PMID 30559816